CLINICAL TRIAL: NCT04497883
Title: A Phase 1, Open-label, Randomized, Cross-over Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of Maribavir Administered in Healthy Japanese Subjects Compared With Matched, Healthy, Non-Hispanic, Caucasian Subjects and to Assess Dose-Proportionality of 3 Doses of Maribavir in the Japanese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of Maribavir Administered in Healthy Japanese Participants Compared With Matched, Healthy, Non-Hispanic, Caucasian Participants and to Assess Dose-Proportionality of 3 Doses of Maribavir in Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-1020
Record Dates: First submitted 2020-07-07; First posted 2020-08-04 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Non-Hispanic, Caucasian (Experimental): Non-Hispanic, Caucasian group participants will receive 400 milligram (mg) maribavir tablets orally once on Day 1 during treatment period 1.
  Interventions: Drug: Maribavir (400 mg)
- Cohort B: Japanese Descent (Experimental): Japanese descent group participants will receive 400 mg maribavir tablets orally once on Day 1 during treatment period 1 followed by 200 mg or 800 mg maribavir tablets orally once on Day 1 during treatment period 2 followed by 800 mg or 200 mg maribavir tablets orally once on Day 1 during treatment period 3 in cross-over fashion. A washout period of 72 hours will be maintained between treatment period 1, 2, and 3.
  Interventions: Drug: Maribavir (400 mg); Drug: Maribavir (200 mg); Drug: Maribavir (800 mg)

INTERVENTIONS:
Drug: Maribavir (400 mg) — Non-Hispanic, Caucasian group and Japanese descent group participants will receive 400 mg maribavir tablets orally once on Day 1 during treatment period 1.
  Other Names: SHP620; TAK-620
Drug: Maribavir (200 mg) — Japanese descent group participants will receive 200 mg maribavir tablets orally once on Day 1 during treatment period 2 or 3.
  Other Names: SHP620; TAK-620
  Arms: Cohort B: Japanese Descent
Drug: Maribavir (800 mg) — Japanese descent group participants will receive 800 mg maribavir tablets orally once on Day 1 during treatment period 2 or 3.
  Other Names: SHP620; TAK-620
  Arms: Cohort B: Japanese Descent

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK), safety, and tolerability of maribavir administered as a single oral dose in healthy, adult participants of Japanese descent and matched, healthy, adult, non-Hispanic, Caucasian participants. In addition, this study will assess the dose-proportionality of PK of maribavir in healthy, adult participants of Japanese descent.

DETAILED DESCRIPTION:
The study will be conducted in two cohorts, Cohort A and Cohort B. Cohort A consists of 12 participants of Japanese Descent. Cohort B consists of 12 non-Hispanic, Caucasian participants.

For Japanese participants there will be three treatment periods. In Treatment Period 1, they will receive maribavir as a single 400 mg oral dose. In Treatment Periods 2 and 3, all Japanese participants will receive maribavir as a single oral dose of either 200 mg or 800 mg, depending upon randomization assignment. For the non-Hispanic, Caucasian group there will be only one treatment period and they will receive maribavir as a single 400 mg oral dose.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written informed consent/assent as applicable to participate in the study.
* Healthy 18 to 55 years old participants of Japanese descent and non-Hispanic Caucasian origin.
* Healthy participants of Japanese descent must have been born in Japan and must not have lived outside of Japan for greater than (>) 10 years; both parents and all 4 grandparents must be of Japanese origin. Healthy, non-Hispanic, Caucasian participants must have both parents and all 4 grandparents of non-Hispanic, Caucasian origin.
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Hemoglobin for males greater than or equal to (>=) 135.0 gram per liter (g/L) and females >= 120.0 g/L at screening and on Day -1.
* Body mass index (BMI) between 18.5 and 28.0 kilogram per square meter (kg/m^2) inclusive with a body weight > 45 kilograms (kg) (99 pounds [lbs]).
* Ability to swallow a dose of investigational product (IP).

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological, or psychiatric disease, gall bladder removal, or current recurrent disease.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures.
* Known or suspected intolerance or hypersensitivity to maribavir, closely-related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of IP.
* Donation of blood or blood products (e.g. plasma or platelets) within 60 days prior to receiving the first dose of IP.
* Have taken another IP within 30 days or five half-lives of that IP, whichever is greater, prior to the first dose of maribavir.
* Have been enrolled in a clinical study (including vaccine studies) within 30 days prior to the first dose of IP that, in the investigator's opinion, may impact this study.
* Have had any substantial changes in eating habits within 30 days prior to the first dose of IP, as assessed by the investigator.
* Confirmed systolic blood pressure > 139 millimeter of mercury (mmHg) or less than (<) 89 mmHg, and diastolic blood pressure > 89 mmHg or < 49 mmHg.
* Twelve-lead ECG demonstrating QTc > 450 milliseconds (msec).
* Known history of alcohol or other substance abuse, including synthetic cannabinoids within the last year.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day.
* A positive urine test for drugs of abuse, alcohol, or cotinine at screening or on Day -1.
* A positive human immunodeficiency virus (HIV), hepatitis B surface antibody (HBsAg), or hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form (e.g. smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch).
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches.
* Current use of any prescription medication within 30 days of the first dose of IP. Current use of any over the counter medication within 14 days of the first dose of IP.
* Ingestion of known cytochrome P450 (CYP) 3A modulators within 7 days of Day 1, period 1
* History of active or chronic oral/nasal cavity infections, gastroesophageal reflux, asthma treatment with albuterol, zinc supplementation.
* Participants with dry mouth syndrome or burning mouth syndrome or menopausal women suffering from dysgeusia.
* Participants who have acute gastrointestinal (GI) symptoms at screening or admission (e.g. nausea, vomiting, diarrhea, and heartburn).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- PPD Development, LP, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5facfd1e17465c002989a19b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in the United States from 07 Aug 2020 (first participant first visit) to 12 Nov 2020 (last participant last visit).
Pre-assignment Details: A total of 24 participants (12 non-Hispanic Caucasian participants in Cohort A and 12 Japanese participants in Cohort B) were enrolled, randomized and received the study treatment in this study.
Groups:
- Cohort A: Non-Hispanic, Caucasian: Non-Hispanic, Caucasian participants received single dose of 400 milligram (mg) maribavir tablets orally on Day 1 during treatment period 1.
- Cohort B: Japanese Descent: Maribavir 400mg: Japanese descent participants received single oral dose of 400 mg maribavir tablets on Day 1 during treatment period 1.
- Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg: Japanese descent participants who received 400 mg maribavir tablets during treatment period 1 received single dose of 200 mg maribavir tablet orally on Day 1 during treatment period 2 followed by single dose of 800 mg maribavir tablets orally on Day 1 during treatment period 3. A washout period of 72 hours was maintained between treatment period 1, 2, and 3.
- Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg: Japanese descent participants who received 400 mg maribavir tablets during treatment period 1 received single dose of 800 mg maribavir tablets orally on Day 1 during treatment period 2 followed by single dose of 200 mg maribavir tablet orally on Day 1 during treatment period 3. A washout period of 72 hours was maintained between treatment period 1, 2, and 3.
Period: Treatment Period 1 (2 Days)
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent: Maribavir 400mg | Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg | Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg
Started | 12 | 12 | 0 | 0
Completed | 12 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (72 Hours)
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent: Maribavir 400mg | Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg | Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg
Started | 12 | 12 | 0 | 0
Completed | 12 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (2 Days)
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent: Maribavir 400mg | Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg | Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (72 Hours)
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent: Maribavir 400mg | Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg | Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3 (2 Days)
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent: Maribavir 400mg | Cohort B: Japanese Descent: First Maribavir 200 mg Then Maribavir 800 mg | Cohort B: Japanese Descent: First Maribavir 800 mg Then Maribavir 200 mg
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of participants who were administered at least 1 dose of maribavir and had at least 1 post-dose safety assessment.
Groups:
- Cohort A: Non-Hispanic, Caucasian: Non-Hispanic, Caucasian participants received 400 mg maribavir tablets orally once on Day 1 during treatment period 1.
- Cohort B: Japanese Descent: Japanese descent participants received single dose of 400 mg maribavir tablets orally on Day 1 during treatment period 1 followed by single dose of 200 mg or 800 mg maribavir tablets orally on Day 1 during treatment period 2 followed by single dose of 800 mg or 200 mg maribavir tablets orally on Day 1 during treatment period 3 in cross-over fashion. A washout period of 72 hours was maintained between treatment period 1, 2, and 3.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Non-Hispanic, Caucasian | Cohort B: Japanese Descent | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (9.33) | 40.8 (8.92) | 40.0 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 12 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 0 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Maribavir
Description: Cmax of maribavir in plasma were reported.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: The pharmacokinetic (PK) set consisted of participants who received at least 1 dose of maribavir and had evaluable post-dose maribavir PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (mcg/mL)
Groups:
- Cohort A: Maribavir 400 mg: Non-Hispanic, Caucasian participants received single oral dose of 400 mg maribavir tablets on Day 1 during treatment period 1.
- Cohort B: Maribavir 400 mg: Japanese descent participants received single oral dose of 400 mg maribavir tablets on Day 1 during treatment period 1.
- Cohort B: Maribavir 200 mg: Japanese descent participants received single oral dose of 200 mg maribavir tablets on Day 1 during treatment period 2 or 3.
- Cohort B: Maribavir 800 mg: Japanese descent participants received single oral dose of 800 mg maribavir tablets on Day 1 during treatment period 2 or 3.
Arm/Group | Cohort A: Maribavir 400 mg | Cohort B: Maribavir 400 mg | Cohort B: Maribavir 200 mg | Cohort B: Maribavir 800 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Micrograms per milliliter (mcg/mL) | 15.8 (26.6) | 17.4 (27.4) | 9.03 (34.0) | 26.3 (30.7)
Statistical Analysis 1: Comparison: Cohort A: Maribavir 400 mg vs Cohort B: Maribavir 400 mg; The comparison analysis was planned between Cohort A: Maribavir 400 mg and Cohort B: Maribavir 400 mg group participants only; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; ANOVA; % Ratio of Geometric least square means = 110.41, 90% CI 2-sided [91.70 to 132.94]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Maribavir
Description: AUClast of maribavir in plasma were reported.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: The PK set consisted of participants who received at least 1 dose of maribavir and had evaluable post-dose maribavir PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Cohort A: Maribavir 400 mg | Cohort B: Maribavir 400 mg | Cohort B: Maribavir 200 mg | Cohort B: Maribavir 800 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hour*microgram per milliliter (h*mcg/mL) | 75.3 (33.6) | 92.3 (35.3) | 41.3 (40.8) | 183 (40.6)
Statistical Analysis 1: Comparison: Cohort A: Maribavir 400 mg vs Cohort B: Maribavir 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; ANOVA; % Ratio of Geometric least square means = 122.49, 90% CI 2-sided [96.83 to 154.95]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-infinity) of Maribavir
Description: AUC(0-infinity) of maribavir in plasma were reported.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Cohort A: Maribavir 400 mg | Cohort B: Maribavir 400 mg | Cohort B: Maribavir 200 mg | Cohort B: Maribavir 800 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
h*mcg/mL | 77.3 (34.7) | 96.7 (37.1) | 43.0 (42.4) | 195 (43.9)
Statistical Analysis 1: Comparison: Cohort A: Maribavir 400 mg vs Cohort B: Maribavir 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; ANOVA; % Ratio of Geometric least square means = 125.08, 90% CI 2-sided [97.99 to 159.64]

4. Secondary Outcome: Dose Proportionality of Cmax of Maribavir in Japanese Descent Participants
Description: Dose proportionality was assessed using the power model including log-transformed Cmax dependent variable and the log-transformed dose as a fixed effect. Natural log (ln) and 90% confidence interval for the slope are presented.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: The PK set consisted of participants who received at least 1 dose of maribavir and had evaluable post-dose maribavir PK data. Dose proportionality of Cmax of maribavir was planned to be evaluated in Japanese descent participants only.
Measure: Number (90% Confidence Interval); unit: ln (Cmax [mcg/mL])
Groups:
- Cohort B: Japanese Descent: All Japanese descent participants who received single dose of 400 mg maribavir tablets orally on Day 1 during treatment period 1 followed by single dose of 200 mg or 800 mg maribavir tablets orally on Day 1 during treatment period 2 followed by single dose of 800 mg or 200 mg maribavir tablets orally on Day 1 during treatment period 3 in cross-over fashion. A washout period of 72 hours was maintained between treatment period 1, 2, and 3.
Arm/Group | Cohort B: Japanese Descent
Number analyzed (Participants) | 12
ln (Cmax [mcg/mL]) | 0.771 [0.62 to 0.92]

5. Secondary Outcome: Dose Proportionality of AUClast of Maribavir in Japanese Descent Participants
Description: Dose proportionality was assessed using the power model including log-transformed AUClast dependent variable and the log-transformed dose as a fixed effect. ln and 90% confidence interval for the slope are presented.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: The PK set consisted of participants who received at least 1 dose of maribavir and had evaluable post-dose maribavir PK data. Dose proportionality of AUClast of maribavir was planned to be evaluated in Japanese descent participants only.
Measure: Number (90% Confidence Interval); unit: ln (AUClast[h*mcg/mL])
Arm/Group | Cohort B: Japanese Descent
Number analyzed (Participants) | 12
ln (AUClast[h*mcg/mL]) | 1.07 [0.89 to 1.26]

6. Secondary Outcome: Dose Proportionality of AUC0-infinity of Maribavir in Japanese Descent Participants
Description: Dose proportionality was assessed using the power model including log-transformed AUC0-inifinity dependent variable and the log-transformed dose as a fixed effect. ln and 90% confidence interval for the slope are presented.
Time Frame: Day 1 of each treatment period: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, and 24 hours post-dose
Population: The PK set consisted of participants who received at least 1 dose of maribavir and had evaluable post-dose maribavir PK data. Dose proportionality of AUC0-infinity of maribavir was planned to be evaluated in Japanese descent participants only.
Measure: Number (90% Confidence Interval); unit: ln (AUC0-infnity[h*mcg/mL])
Arm/Group | Cohort B: Japanese Descent
Number analyzed (Participants) | 12
ln (AUC0-infnity[h*mcg/mL]) | 1.09 [0.90 to 1.29]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily had a causal relationship with this investigational product (IP) or medicinal product. An SAE was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. A TEAE was any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. Number of Participants with TEAEs and serious TEAEs were reported in both non-Hispanic, Caucasian and Japanese descent participants.
Time Frame: From start of study drug administration to follow-up (up to Day 23)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Maribavir 400 mg | Cohort B: Maribavir 400 mg | Cohort B: Maribavir 200 mg | Cohort B: Maribavir 800 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Participants with TEAEs | 4 | 2 | 1 | 0
  Participants with serious TEAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration to follow-up (up to Day 23)
Arm/Group | Cohort A: Maribavir 400 mg | Cohort B: Maribavir 400 mg | Cohort B: Maribavir 200 mg | Cohort B: Maribavir 800 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 2/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Maribavir 400 mg (N=12) | Cohort B: Maribavir 400 mg (N=12) | Cohort B: Maribavir 200 mg (N=12) | Cohort B: Maribavir 800 mg (N=12)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT04497883/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT04497883/SAP_001.pdf